CLINICAL TRIAL: NCT06943677
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TQB3019 Capsules in Subjects With Advanced Malignant Tumors
Brief Title: A Clinical Trial on the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TQB3019 Capsule in Subjects With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3019-I-01
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignant Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3019 capsules (Experimental): Single or continuous administration, 50-600 mg each time TQB3019 capsule is taken orally once a day on an empty stomach, and each cycle is 28 days.
  Interventions: Drug: TQB3019 capsules

INTERVENTIONS:
Drug: TQB3019 capsules — TQB3019 capsule is a targeted protein degrader

SUMMARY:
The trial was divided into two phases: dose escalation and dose expansion. The dosing regimens were single-dose study and continuous dosing study. A single-center, open, non-randomized, single-arm clinical trial design was adopted. Subjects with advanced malignant tumors were selected to take TQB3019 capsules orally to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of TQB3019 capsules.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined the study, signed informed consent form, and with good compliance.
* ≥18 years old; Eastern Cooperative Oncology Group (ECOG) physical status: 0-2; at least 3 months expected survival period.
* Clearly diagnosed recurrent / refractory hematological tumors that meet the World Health Organization (WHO) definition;
* At least 1 measurable lesion for efficacy evaluation.
* The function of main organs is normal.
* Female patients of childbearing age should agree to use contraceptive measures during the study period and for at least 6 months after study is stopped; a negative serum pregnancy test within 7 days prior to study enrollment and must be non-lactating subjects; male patients should agree to use contraception during the study period and for at least 6 months after study is stopped.

Exclusion Criteria:

* Patients has had or is currently having other malignant tumors within 3 years. The following two conditions can be included in the group: other malignant tumors treated with a single operation to achieved 5 consecutive years of disease free survival (DFS)s. Cured cervical carcinoma in situ, non-melanoma skin cancer, nasopharyngeal carcinoma and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)].
* Subjects with central nervous system aggression (CNS);
* Received allogeneic hematopoietic stem cell transplantation (allo-HSCT) or had active graft-versus-host disease (GVHD) requiring immunosuppressive therapy within 12 months before the first dose;
* Multiple factors that affect the absorption of oral medications (e.g., inability to swallow, chronic diarrhea, and intestinal obstruction);
* Unrelieved toxicity of ≥CTC AE grade 1 due to any previous treatment, excluding alopecia and fatigue;
* Major surgical treatment, open biopsy, and significant traumatic injury were received within 28 days before the start of study treatment.
* The presence of active or uncontrolled primary autoimmune cytopenia, including autoimmune hemolytic anemia (AIHA) and primary immune thrombocytopenia (ITP);
* Patients with evidence or history of bleeding constitution; Or any bleeding event (such as gastrointestinal bleeding) greater than or equal to CTC AE level 3 within 4 weeks before the first medication;
* Subjects had an arteriovenous thrombosis event within 6 months.
* Subjects have history of psychotropic substance abuse and are unable to abstain or have mental disorders;
* Subjects with any severe and/or uncontrolled disease.
* Within 2 weeks before the first treatment, the subjects had received proprietary Chinese medicines with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions;
* Previously received treatment with drugs similar to TQB3019 capsules;
* Uncontrolled pleural effusion, pericardial effusion, or ascites that still require repeated drainage (investigator judgment)
* Study treatment related: subjects received live or messenger RNA (mRNA) vaccines within 4 weeks before the first treatment or were scheduled to receive live or mRNA vaccines during the study;
* Participated in clinical trials of other antitumor drugs within 4 weeks before the first treatment;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered unsuitable for enrollment for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (Each cycle is 28 days)
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI Common Terminology Criteria for Adverse Events(CTCAE) version5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred from first medication to the end of the first treatment cycle.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (Each cycle is 28 days)
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose (RP2D) | Baseline up to 24 months
  DLT describes side effects of a drug or other treatment that are serious enough to evaluate RP2D of TQB3019 capsules in adult patients with Advanced Malignant Cancer.
Maximum assessed dose (MAD) | Baseline up to 24 months
  Recommendations made by the investigator and sponsor based on clinical safety, efficacy, pharmacokinetic, and pharmacodynamic data will be considered the highest dose level to complete dose exploration in the absence of an MTD
Adverse events (AEs) | From the time the subject receives TQB3019 to 28 days after the last dose or until the start of other anti-tumor treatment (whichever occurs first, up to approximately 3 years)
  The occurrence of all adverse events (AEs)
Serious adverse events (SAEs) | From the time the subject receives TQB3019 to 28 days after the last dose or until the start of other anti-tumor treatment (whichever occurs first, up to approximately 3 years)
  The occurrence of all serious adverse events (SAEs) .
Abnormal incidence of laboratory test indicators | From the time the subject receives TQB3019 to 28 days after the last dose or until the start of other anti-tumor treatment (whichever occurs first, up to approximately 3 years)
  Incidence and severity of abnormal laboratory values
Overall response rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, up to approximately 3 years
  The proportion of subjects with best response of Complete Response (CR), Partial Response (PR), Partial Response with Lymphocytosis (PR-L), Very Good Partial Response (VGPR), and Minimal Response (MR).

SECONDARY OUTCOMES:
Tmax | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle 1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  Time to Reach the Maximum Plasma Concentration.
Cmax | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  Cmax is the maximum plasma concentration of TQB3019.
Elimination half-life (t1/2) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  To evaluate the Elimination half-life (t1/2) after oral dose of TQB3019 capsules to subjects.
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  To characterize the pharmacokinetics of TQB3019 by assessment of area under the plasma concentration time curve from the first dose to a certain time.
Apparent clearance (CL/F) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body..
Apparent volume of distribution (Vd/F) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  Apparent volume of distribution of the TQB3019 in plasma.
Minimum concentration (Cmin) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  Minimum observed concentration (Cmin) of TQB3019
Bruton's tyrosine kinase (BTK) protein levels | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  BTK protein levels in peripheral blood mononuclear cells (PMBCs)
Complete Remission Rate (CRR) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  The proportion of tumors that have a complete response after treatment.
Disease Control Rate (DCR) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  The percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a cancer treatment in clinical trials.
Duration of Response (DOR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100weeks
  The time from the date of first documentation of a CR or PR or PD to the date of first documentation of tumor progression.
Progression Free Survival (PFS) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  The time from the first dose to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first
Overall Survival (OS) | Single Day1/First dose: pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 hours post dose Cycle1 Day 8, 15, 28: pre-dose; 0.5, 1, 2, 4, 6, 8, 12, 24 hours at days 28 post dose, each cycle is 28 days
  the time from start of study treatment to date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Cancer Institute & Hospital.Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Heze Municipal Hospital, Heze, Shandong
  - The Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Affiliated Hospital of North sichuan Medical college, Nanchong, Sichuan
  - TianJin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality
  - Institute of Hematology ＆Blood Diseases Hospital,Chinese Academy of Medical Sciences ＆Peking Union Medical College, Tianjin, Tianjin Municipality